CLINICAL TRIAL: NCT07078487
Title: Implications of Paced Heart Rate on Central Blood Pressure in Sick Sinus Syndrome Patients With Hypertension: a Randomised Crossover Study
Brief Title: Effect of Paced HR on Central BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Priit Kampus, Associate Professor Priit Kampus, University of Tartu
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 299/T-22
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Sick Sinus Syndrome; Hypertension
Keywords: heart rate; hypertension; sick sinus syndrome; arterial pressure; pulse wave analysis
MeSH Terms: conditions — Sick Sinus Syndrome; Hypertension | interventions — Defibrillators

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Slow" arm (Experimental): Pacemaker base rate set at 55 bpm
  Interventions: Device: Pacemaker and defibrillator
- "Fast" arm (Experimental): Pacemaker base rate set at 75 bpm
  Interventions: Device: Pacemaker and defibrillator

INTERVENTIONS:
Device: Pacemaker and defibrillator — Setting the pacemaker base rate at a pre-defined base rate

SUMMARY:
Central (aortic) blood pressure predicts heart, brain and kidney complications more reliably than the usual peripherally measured blood pressure. Heart rate has a strong and sometimes counter-intuitive influence on central blood pressure. Pacemakers implanted due to sick sinus syndrome (SSS) are typically programmed anywhere between 55-75 beats per minute (bpm), yet it is unclear which rate gives hypertensive pacemaker recipients the most favourable central hemodynamics.

This single-center, randomized, single-blind, two-period cross-over trial will enrol 20 adults (18-80 years) who already carry a dual-chamber pacemaker for SSS, are in sinus rhythm, and have medication-controlled arterial hypertension. Each participant will complete two eight-week pacing periods in random order:

* "Slow" period - pacemaker lower-rate set to 55 bpm.
* "Fast" period - pacemaker lower-rate set to 75 bpm.

A two-week wash-out at the device's usual settings separates the periods. At baseline and after each intervention the team will perform non-invasive pulse-wave analysis (SphygmoCor XCEL) to obtain central systolic blood pressure (primary endpoint) and arterial stiffness indices such as augmentation index and pulse-wave velocity (secondary endpoints). Pacemaker function, symptoms and safety events are reviewed at every visit; settings can be adjusted by ±5 bpm if troublesome symptoms occur.

The study will provide the first long-term evidence on how fixed pacing rates modulate central blood pressure in real-world SSS patients with hypertension, potentially guiding clinicians toward the optimal programming strategy.

DETAILED DESCRIPTION:
Scientific background and rationale Arterial hypertension remains the leading modifiable contributor to cardiovascular morbidity. Unlike brachial pressure, central (aortic) systolic pressure directly loads the left ventricle and cerebral and renal arteries. Epidemiological data show that central pressure is more closely associated with left-ventricular hypertrophy, carotid atherosclerosis and clinical events than peripheral pressure. Heart rate (HR) alters the timing of pulse-wave reflections and can therefore change central pressure in ways that are not apparent from arm-cuff readings.

Pharmacological HR reduction (e.g., ivabradine) has been shown to raise central systolic pressure even while lowering brachial pressure, whereas β-blockers exert mixed HR-dependent and HR-independent effects. In acute pacing studies, lowering HR from 80 bpm to ~60 bpm reduced brachial pressure but left central pressure unchanged; allowing HR to fall to ~50 bpm sometimes lowered or sometimes raised central pressure depending on study design. No prospective trial has tested whether a chronically lower versus higher pacemaker rate produces a durable difference in central hemodynamics in patients who require pacing for SSS.

Objectives Primary: Compare clinic-measured central systolic blood pressure after 8 weeks of pacing at 55 bpm versus 75 bpm.

Secondary: Compare additional central hemodynamic indices (augmentation index, pulse pressure amplification, carotid-femoral pulse-wave velocity), brachial blood pressure, and frequency of pacing-related symptoms and atrial arrhythmias between the two settings.

Study design

* Single-center, randomized, single-blind, cross-over.
* Two 8-week intervention periods separated by a 2-week wash-out.
* Allocation ratio 1:1, block randomization, concealed in sequentially numbered opaque envelopes prepared by an independent statistician.

Visit schedule

T-2 (pre-screen) → T-1 (final screen + baseline PWA) → T0 (randomization) → T1 (programming of first rate) → 8 weeks → F1 (end-of-period assessments, device reset) → 2-week wash-out → T2 (second baseline) → program second rate → 8 weeks → F2 (final assessments, device returned to pre-study settings). Total participation ≈20 weeks.

Participants Inclusion

1. Age 18-80 years.
2. Dual-chamber pacemaker implanted ≥3 months for SSS.
3. Sinus rhythm; atrial pacing >80%, ventricular pacing <3% since last device check.
4. Medication-treated primary hypertension with clinic BP < 140/90 mmHg and home BP < 135/85 mmHg.
5. Able to provide informed consent and comply with procedures. Exclusion (abridged)

   * Significant AV block, paced QRS ≥ 130 ms, >3 antihypertensives, digoxin or class Ic/III/IV antiarrhythmics, frequent atrial tachyarrhythmia (>3% AMS episodes), coronary intervention on >1 vessel, LVEF ≤ 40%, CRT or ICD, significant valvular disease, congenital heart disease, BMI ≥ 35 kg/m², diabetes with complications or on insulin, advanced renal, hepatic or pulmonary disease, systemic inflammatory disease, malignancy under recent active therapy, pregnancy or lactation, substance misuse, or inability to complete follow-up.

Interventions Pacemaker lower-rate limit is set to either 55 bpm or 75 bpm using a Merlin™ Patient Care programmer (Abbott/St Jude Medical). All other device parameters remain unchanged unless clinically indicated. If intolerable palpitations, dizziness or dyspnoea occur, HR may be adjusted by ±5 bpm within protocol limits; the participant may continue.

Sample size and statistics The initial 20-patient cohort (2020-2022) showed a within-person SD of 5 mmHg for central systolic BP. Detecting a 3 mmHg difference with 80% power at α = 0.05 in a cross-over design requires 38 completed participants; 20 additional individuals will therefore be recruited (total = 40) to allow for 5% attrition. Analysis will follow an intention-to-treat principle.

Data collection methods

Pulse-wave analysis: SphygmoCor XCEL (AtCor Medical) brachial cuff acquisition with generalized transfer function yields central waveforms. Carotid-femoral pulse-wave velocity is obtained by simultaneous carotid tonometry and femoral cuff recording with surface tape measurement of path length. Standardized seated brachial BP is averaged from triplicate readings. Home BP is logged using a validated oscillometric device. Device diagnostics supply pacing percentages and arrhythmia burden.

Safety, monitoring and ethics All procedures mirror routine pacemaker follow-up except for deliberate lower-rate reprogramming, which falls within the accepted clinical range (55-75 bpm). The prior 20-participant phase recorded two episodes of atrial fibrillation requiring treatment and no serious device malfunctions. Adverse events will be reported to the ethics committee within 15 days. The study complies with the Declaration of Helsinki, EU GDPR and ICH-GCP. Data are pseudonymised; records are stored on secure servers for 10 years, after which they are destroyed. The University of Tartu Human Research Ethics Committee has approved the protocol (initial approval 299/T-22, renewed 2025).

Dissemination Results will be submitted to a peer-reviewed cardiovascular journal, presented at international cardiology conferences.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Dual-chamber pacemaker implanted ≥3 months for SSS.
3. Sinus rhythm; atrial pacing >80%, ventricular pacing <3% since last device check.
4. Medication-treated primary hypertension with clinic BP < 140/90 mmHg and home BP < 135/85 mmHg.
5. Able to provide informed consent and comply with procedures.

Exclusion Criteria:

Significant AV block, paced QRS ≥ 130 ms, >3 antihypertensives, digoxin or class Ic/III/IV antiarrhythmics, frequent atrial tachyarrhythmia (>3% AMS episodes), coronary intervention on >1 vessel, LVEF ≤ 40%, CRT or ICD, significant valvular disease, congenital heart disease, BMI ≥ 35 kg/m², diabetes with complications or on insulin, advanced renal, hepatic or pulmonary disease, systemic inflammatory disease, malignancy under recent active therapy, pregnancy or lactation, substance misuse, or inability to complete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Central systolic blood pressure | After each 8-week intervention period (at week 8 and week 18 of study participation)
  Central (aortic) systolic blood pressure measured non-invasively using pulse wave analysis (SphygmoCor XCEL) with brachial cuff acquisition and generalized transfer function to derive central waveforms. Measurements taken in standardized seated position in clinical setting.

SECONDARY OUTCOMES:
Central diastolic blood pressure | After each 8-week intervention period (at week 8 and week 18 of study participation)
  Central (aortic) diastolic blood pressure measured non-invasively using pulse wave analysis (SphygmoCor XCEL) with brachial cuff acquisition and generalized transfer function to derive central waveforms.
Augmentation index | After each 8-week intervention period (at week 8 and week 18 of study participation)
  Augmentation index derived from central pulse wave analysis measuring the contribution of reflected waves to central systolic pressure, expressed as percentage increase in central systolic pressure due to wave reflection.
Pulse wave velocity | After each 8-week intervention period (at week 8 and week 18 of study participation)
  Carotid-femoral pulse wave velocity measured using simultaneous carotid tonometry and femoral cuff recording with surface measurement of path length, indicating arterial stiffness.
Brachial blood pressure | After each 8-week intervention period (at week 8 and week 18 of study participation)
  Peripheral (brachial) systolic and diastolic blood pressure measured using standardized seated position with triplicate readings averaged, measured using validated oscillometric device.
Pulse pressure amplification | After each 8-week intervention period (at week 8 and week 18 of study participation)
  Ratio of peripheral to central pulse pressure derived from non-invasive pulse wave analysis (SphygmoCor XCEL), reflecting amplification of the pressure wave between the aorta and brachial artery.

CONTACTS AND LOCATIONS:
Locations (1):
- North Estonia Medical Centre, Tallinn, Harju, Estonia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hashimoto J. Pulse pressure amplification as a hemodynamic predictor of cardiovascular disease. Hypertens Res. 2024 Nov;47(11):3270-3272. doi: 10.1038/s41440-024-01880-8. Epub 2024 Sep 11. No abstract available. PMID 39261706
- [Background] Fong DT, Yam KY, Chu VW, Cheung RT, Chan KM. Upper limb muscle fatigue during prolonged Boccia games with underarm throwing technique. Sports Biomech. 2012 Nov;11(4):441-51. doi: 10.1080/14763141.2012.699977. PMID 23259234
- [Background] Ikeda S, Shinohara K, Enzan N, Matsushima S, Tohyama T, Funakoshi K, Kishimoto J, Itoh H, Komuro I, Tsutsui H. A higher resting heart rate is associated with cardiovascular event risk in patients with type 2 diabetes mellitus without known cardiovascular disease. Hypertens Res. 2023 May;46(5):1090-1099. doi: 10.1038/s41440-023-01178-1. Epub 2023 Jan 27. PMID 36707715
- [Background] Fox K, Borer JS, Camm AJ, Danchin N, Ferrari R, Lopez Sendon JL, Steg PG, Tardif JC, Tavazzi L, Tendera M; Heart Rate Working Group. Resting heart rate in cardiovascular disease. J Am Coll Cardiol. 2007 Aug 28;50(9):823-30. doi: 10.1016/j.jacc.2007.04.079. Epub 2007 Aug 13. PMID 17719466